CLINICAL TRIAL: NCT03627364
Title: Analysis of Electrophysiological Markers for Sensorimotor Recovery in Post Stroke Patients
Brief Title: Analisys of Cortical Excitability and Motor Function of Post Stroke Patients
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Principal investigator, Universidade Federal de Pernambuco
Other Study IDs: motor function_stroke
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Stroke; Motor Function; Cortical Excitability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post stroke patients: will be submitted to a single session to obtain the normal neurophysiological and behavioral endpoints and thus compare with those obtained in healthy individuals.
- Control group: will be submitted to a single session to obtain the normal neurophysiological and behavioral endpoints and thus compare with those obtained in post stroke patients.

SUMMARY:
Healthy individuals, after reading and signing the free and informed consent will be submitted to a single session to obtain the normal neurophysiological measures and thus compare with those obtained in individuals with PD. Healthy and post stroke patients will be submitted to a neurophysiological evaluation through transcranial magnetic stimulation (TMS) and electroencephalography (EEG). The post stroke patients will also performed the evaluation trought the fugl meyer scale.

DETAILED DESCRIPTION:
Fugl Meyer assesment is used to measure motor control recovery. It is a 226 point scoring system that includes the following sessions: range of motion, pain, sensation,motor function of upper and lower limbs, balance, coordination and velocity. The investigators will aplly only two sessions: upper limb motor function and coordination/velocity, these sessions totalize 66 points.

Cortical excitability level it will be evaluated through single pulse transcranial magnetic stimulation paradigms (Neurosoft, Russia). Initially, rest motor threshold (RMT) will be determined by finding the lowest stimulator output that elicit motor evoked potential (MEP) around 50 μV (TMS Motor Threshold Assessment Tool -MTAT 2.0 - USA). For RMT measure, a figure-eight coil connected to the magnetic stimulator held manually at 45 degrees from the midline, will be placed over the right primary motor cortex of lesioned and non lesioned hemisphere (C3 and/or C4 - 10/20 System). After, motor evoked potential will be evaluet by 20 pulses firing with 120% of RMT.

EEG Patients will perform an assessment of brain activity through the EEG. Initially, patients will be placed seated in a chair at 90cm in front of a computer. Then, the equipment will be assembled, the points according to the 10-20 marking system will be identified: Cz, C3, C4, F3, F4, P3, P4, Fz and Pz.

The protocol will follow the sequence of six consecutive moments (1 minute each) to monitor the patient's brain activity through Neuro Spectrum software:

1. 1st minute: REST: the patient will be relaxed, at rest, without any communication and with eyes open;
2. 2nd minute: OBSERVE - the patient will observe the video of the movement hand to mouth;
3. 3rd minute: EXECUTION - the patient will reproduce the movement of the video with healthy limb (post stroke patient)/ dominant hand (healthy);
4. 4th minute: IMAGINATION - the patient will imagine the previous movement;
5. 5th minute: EXECUTION - the patient will reproduce the movement of the video with a paretic limb (post stroke patient)/ non dominant hand (healthy);
6. 6th minute: IMAGINATION - the patient will imagine the previous movement;

ELIGIBILITY:
Inclusion Criteria:

* Post stroke patients

  • Primary or recurrent, ischemic or hemorrhagic stroke, confirmed by computed tomography or magnetic resonance imaging
* Chronic Stroke (> 3 months)

  * Sensorimotor sequelae in an upper limb due to stroke
  * Score ≥ 18 at Folstein Mini Mental State Examination Healthy Subjects
  * Ages: 40 years or greater
  * Gender: Both
  * Subjects who do not have self-report of neurological or articular disorder

Exclusion Criteria:

* Post stroke patients

  * Prior neurological diseases
  * Multiple brain lesions
  * Metal implant in the skull and face
  * Pacemaker
  * History of seizures
  * Epilepsy
  * Pregnancy
  * Hemodynamic instability
  * Traumatic orthopedic injuries of upper limb that compromise the function
  * Altered medication for less than 3 months or who underwent botulinum toxin for less than 6 months
  * Performing physical therapy elsewhere during the period of intervention Healthy Subjects
  * Pregnant women;
  * Pacemaker;
  * History of seizures;
  * Metallic implants in the head;
  * Patients with clinical evidence of brain injuries;
  * Chronic pain associated to other diseases;
  * Use of neuroleptic medications
  * Individuals with other neurological disorders, postural hypotension, vestibular, visual, cardiovascular or musculoskeletal disorders that affect the performance of the proposed tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population study was composite for patients post-stroke with auditory major that 3 months and found in the eligibility criteria. In addition, it will rely on babies with health or neurological disorders.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
sensory-motor recovery level | baseline
  Fugl Meyer assesment of paretic upper limb motor function is used to measure motor control recovery. It is a 226 point scoring system that includes the following sessions: range of motion, pain, sensation,motor function of upper and lower limbs, balance, coordination and velocity. We will aplly only two sessions: upper limb motor function and coordination/velocity, these sessions totalize 66 points

SECONDARY OUTCOMES:
Cortical excitabilit level | baseline
  it will be evaluated through single pulse transcranial magnetic stimulation paradigms (Neurosoft, Russia). Initially, rest motor threshold (RMT) will be determined by finding the lowest stimulator output that elicit motor evoked potential (MEP) around 50 μV (TMS Motor Threshold Assessment Tool -MTAT 2.0 - USA). For RMT measure, a figure-eight coil connected to the magnetic stimulator held manually at 45 degrees from the midline, will be placed over the right primary motor cortex of lesioned and non lesioned hemisphere (C3 and/or C4 - 10/20 System). After, motor evoked potential will be evaluet by 20 pulses firing with 120% of RMT
level of cortical electrical activity | baseline
  Patients will perform an assessment of brain activity through the EEG. Initially, patients will be placed seated in a chair at 90cm in front of a computer. Then, the equipment will be assembled, the points according to the 10-20 marking system will be identified: Cz, C3, C4, F3, F4, P3, P4, Fz and Pz.
  The protocol will follow the sequence of six consecutive moments (1 minute each) to monitor the patient's brain activity through Neuro Spectrum software.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Applied Neuroscience Laboratory, Universidade Federal de Pernambuco, Recife, Pernambuco
  - Applied Neuroscience Laboratory, Recife, Pernambuco

IPD SHARING:
Plan to Share IPD: No